CLINICAL TRIAL: NCT04662359
Title: Ultrasound to Enhance Treat-to-Target in Rheumatoid Arthritis: A Cross-sectional Study
Brief Title: Ultrasound Efficacy in Moderate Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Michael George, MD, MSCE, Assistant Professor, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 844254
Record Dates: First submitted 2020-11-30; First posted 2020-12-10 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Ultrasound
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: This single-arm pilot interventional study will evaluate the potential for ultrasound to improve disease activity assessments for patients with rheumatoid arthritis with clinical scores indicating moderate or high disease activity. Patient facing measures including the Routine Assessment of Patient Index Data (RAPID)3 and the Clinical Disease Activity (CDAI) will be used to determine patient disease activity, as well as whether patients are eligible for the study. The investigators will also collect inflammatory marker levels (including C-reactive protein) and ultrasound assessment to determine severity of illness and for physicians to determine treatment recommendations. Additional patient information will be obtained via chart reviews, and providers will complete pre- and post-ultrasound assessments of the patients.
Masking Description: All patients will receive the ultrasound assessment, so there is no need for masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ultrasound Assessment of Rheumatoid Arthritis Severity (Other): All patients will receive an ultrasound scan to assess the severity of their arthritis. This scan will then be placed in their medical record to allow their rheumatologist to utilize the scan when making treatment recommendations.
  Interventions: Diagnostic Test: Ultrasound Assessment

INTERVENTIONS:
Diagnostic Test: Ultrasound Assessment — Patients will undergo an ultrasound scan to assess the severity of their rheumatoid arthritis.

SUMMARY:
The objectives of this research study are to determine the frequency of low synovitis scores by ultrasound in patients with Rheumatoid Arthritis in moderate or high disease activity and to compare physician treatment recommendations for patients before versus after receiving ultrasound results. Participants will answer questionnaires about their disease activity and complete a musculoskeletal ultrasound in accordance with the study procedures.

DETAILED DESCRIPTION:
The purpose of this research study is to determine whether ultrasound technology can improve treatment decisions for patients with rheumatoid arthritis who have elevated disease activity scores. To do so, the investigators will be evaluating rheumatoid arthritis patients with moderate to high disease activity and how ultrasound scans can reveal any new information about the severity of their arthritis. Patients will answer questionnaires to gauge their disease activity as well as the depression, fatigue, and pain they experience as a result of their arthritis. The patients will then undergo an ultrasound examination to evaluate their synovitis levels, which will then be made available to their physician. Physicians will be asked about their disease activity assessments and treatment recommendations before and after ultrasounds are performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the American College of Rheumatology's 2010 criteria for rheumatoid arthritis. They must be undergoing treatment with a disease-modifying anti-rheumatic drug, and their Clinical Disease Activity Index (CDAI) must be greater than 10 while their swollen joint count must be less than or equal to two.

Exclusion Criteria:

* Patients with evidence of large joint (knee, hip, shoulder, elbow) disease activity, including warmth and swelling, and patients who have had a joint MRI or musculoskeletal ultrasound in the past 3 months will not be eligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael George, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasound Assessment of Rheumatoid Arthritis Severity
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ultrasound Assessment of Rheumatoid Arthritis Severity
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
Rheumatoid arthritis disease duration [Mean (Standard Deviation); unit: years] | 14 (12)

OUTCOME MEASURES:

1. Primary Outcome: Low Synovitis Scores
Description: The primary outcome variable is the proportion of patients with low synovitis scores, which will be determined by the ultrasound assessment. These scores will also be compared to other measures of disease activity. The investigators will be using the EULAR-OMERACT (European League Against Rheumatism - Outcome Measures in Rheumatology) combined scoring system for grading synovitis in rheumatoid arthritis. Each joint is scored from 0-3 with higher scores indicating higher inflammatory activity. Patients with scores of 1 or below in all measured joints are considered to have low synovitis scores.
Time Frame: The outcome is assessed at the time of ultrasound
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound Assessment of Rheumatoid Arthritis Severity
Number analyzed (Participants) | 18
Participants | 1

2. Secondary Outcome: Treatment Recommendations
Description: The secondary outcome will be the number of patients for which the ultrasound information changed the treatment recommendation of the clinical provider.
Time Frame: This measure is assessed after ultrasound results are available (1-2 weeks after ultrasound is performed) based on provider survey
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound Assessment of Rheumatoid Arthritis Severity
Number analyzed (Participants) | 18
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of enrollment through completion of ultrasound (within 3 months)
Description: standard definitions used
Arm/Group | Ultrasound Assessment of Rheumatoid Arthritis Severity
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT04662359/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT04662359/ICF_001.pdf